CLINICAL TRIAL: NCT02774395
Title: Endometrial Cancer and Fractalkine-receptor Axis of Fractalkine
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Other Study IDs: 15-AOI-09
Record Dates: First submitted 2016-05-10; First posted 2016-05-17 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — endometrioid adenocarcinoma and healthy endometrioid (obtain after hysterectomia)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- endometrioid adenocarcinoma grade I
- endometrioid adenocarcinoma grade II
- endometrioid adenocarcinoma garde III
- healthy endometrioid: obtain after hysterectomia provided for

SUMMARY:
The endometrial cancers are among the most common malignancies in postmenopausal women with an incidence on the rise. It is most often a endometrioid adenocarcinoma (grade I, II, III). Other histological types are represented mainly by the clear cell carcinoma, papillary serous carcinoma, the carcinosarcoma. The main risk factors for endometrial cancer are age, obesity, diabetes, hypertension, hormone replacement therapy with estrogen and tamoxifen.

Endometrial hyperplasia usually precedes endometrial cancer is classified by degree of cytologic atypia. Tumor grade quantifies the degree of differentiation and significantly influences the prognosis. Most research has been applied to define the role of estrogen in these cancers, however an accumulation of data indicate that the general process of tumorigenesis is closely related to immune and inflammatory microenvironment of the tumor. In fact, the microenvironment may be seen as a prognostic parameter of tumors or even predictive of therapeutic response.

Recognized as the key molecules responsible for leukocyte recruitment into the tissues, the chemokine-receptor pairs are key players in the immune response, including the anti-tumor immune response but also the inflammatory response. The chemokine-receptor pairs are also involved in many other basic processes such as proliferation, survival or cell death.

The objective of this study was to evaluate the prognostic value of the expression of the chemokine fractalkine (FKN) and its receptor CX3CR1 for the development of endometrioid adenocarcinomas.

Chemokine FKN has the particularity to exist in two forms, a soluble (FKNs), like all chemokines and membrane form (FKNm). The FKNs, resulting from proteolytic cleavage of the FKNm, is provided with chémoattractantes properties. FKNm the present adhesion molecule properties.

The role of FKN in cancer biology is complex.

To date, the role of FKN in endometrial cancer has not been reported. Similarly, the precise role of FKN in the physiology of the endometrium is unknown.

Nevertheless, fractalkine is one of the most expressed in endometrial chemokines. The expression of FKN and its CX3CR1 receptor is detected in the endometrium at all stages of the menstrual cycle. The respective levels of expression of each are fluctuating and largely dependent on the cycle of stage suggesting a possible control by estrogen and progesterone control described elsewhere ovarian level and endothelial. The cells of the endometrial glandular epithelium, macrophages, neutrophils and NK cells infiltrated in this tissue as well as the endothelial cells of blood vessels express FKN. Interestingly, all the cells mentioned above express CX3CR1, except for NK cells and unlike most tissues, the CD8 cells, present in the endometrium, do not express CX3CR1.

In addition, the strongest expression of FKN and CX3CR1 cells by endometrial epithelial coincides with the maximum activity of the glandular epithelium suggesting a possible autocrine loop promoting cell proliferation of the endometrium. Concurrently with the peak of fractalkine, an accumulation of monocytes / macrophages and neutrophils is observed in the endometrium. It appears, moreover, that the balance between the soluble and membrane forms of FKN is important for positioning, infiltration and activity of immune cells within the endometrium.

Current knowledge on the involvement of FKN / CX3CR1 axis in the physiology of the endometrium, although incomplete, point unequivocally the potential role of this ligand pair / receptor in the physiology of the tissue and also suggest that a malfunction of this axis could easily cause various diseases.

Chronic inflammation of a tissue, largely dependent on macrophage infiltration rate, generally represents the tumor development. The endometrium is subjected to physiologically cyclic and regular inflammatory episodes, mirrors for the expression of chemokines and leukocyte infiltration. However, prolonged leukocyte infiltration establishing chronic or prolonged inflammation of the endometrium could help shape a favorable microenvironment in tumor development. Curiously, the axis FKN / CX3CR1 is involved in the development of several inflammatory diseases, including obesity and diabetes are also risk factors for endometrial cancer.

A change in the expression of FKN and / or CX3CR1 is potentially capable of altering the inflammatory physiological cycle of the endometrium and therefore likely to be an element to consider in the evaluation of cancer risk factors of the endometrium.

The assumption is that the FKN / CX3CR1 couple could intervene in the pathophysiology of endometrioid adenocarcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from endometrial hypertrophy or endometrial cancer

Exclusion Criteria:

* no

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from endometrial hypertrophy or endometrial cancer
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
expression rate of FKN | 12 months
expression rate of CX3CR1 | 12 months
expression rate of the couple FKN / CX3CR1 | 12 months
  relationship between the expression levels of the couple FKN / CX3CR1

SECONDARY OUTCOMES:
infiltration rate of certain leukocyte populations | 12 months
expression rate of estrogen receptor | 12 months
expression rate of progesterone hormones | 12 months
expression rate of mitotic index or tumor grade | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No